CLINICAL TRIAL: NCT00037570
Title: A Randomized Study of the Effect of Intravenous Pantoprazole on Gastric pH After Successful Hemostasis in Patients With Bleeding Peptic Ulcer
Brief Title: Study Evaluating Pantoprazole in Peptic Ulcer Hemorrhage
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Purpose: Prevention
Other Study IDs: 3001K2-201
Record Dates: First submitted 2002-05-17; First posted 2002-05-20 (Estimated); Last update posted 2013-02-08 (Estimated); Status verified 2013-02

CONDITIONS: Peptic Ulcer Hemorrhage
Keywords: Peptic; Ulcer; Hemorrhage
MeSH Terms: conditions — Peptic Ulcer Hemorrhage; Ulcer; Hemorrhage | interventions — Pantoprazole

INTERVENTIONS:
Drug: Pantoprazole

SUMMARY:
This is a multicenter, randomized, double-blind, parallel-group, dose-ranging, comparator-controlled study of the effect of pantoprazole on intragastric pH after successful endoscopic hemostasis in hospitalized patients. Patients will receive either intravenous pantoprazole (one of two regimens) or ranitidine (the comparator) within 2 hours of successful hemostasis and administration will continue for 72 hours after hemostasis.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be men or nonpregnant women at least 18 years of age
* Patients who present with a gastric or duodenal ulcer (major dimension of the ulcer must be ≥ 5 mm and ≤ 20 mm) with endoscopic appearance of spurting, oozing, or nonbleeding visible vessel (NBVV) Patients presenting with adherent protruding clot are eligible if, after removal of the clot by irrigation, the underlying lesion is classified as spurting, oozing or a NBVV. Patients with an actively bleeding ulcer or a NBVV within a hiatal hernia are eligible if the ulcer is located below the Z-line)

Exclusion Criteria:

* Patients with ulcer appearance of clean base (non-oozing, non-spurting) or flat pigmented spot; adherent clots not removed by irrigation
* Patients presenting with active bleeding and/or NBVV at 2 or more separate sites
* Patients with any severe concomitant diseases, eg, end-stage liver or renal disease, or unstable cardiovascular, pulmonary, renal, hepatic, or gastrointestinal diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2000-11; Primary Completion 2002-02 (Actual); Study Completion 2002-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, MD, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (6):
- United States (6):
  - Los Angeles, California
  - San Diego, California
  - Cincinnati, Ohio
  - Philadelphia, Pennsylvania
  - Houston, Texas
  - Norfolk, Virginia